CLINICAL TRIAL: NCT00386334
Title: A Long-Term Safety and Efficacy Study of Eszopiclone in Elderly Subjects With Primary Chronic Insomnia
Brief Title: A Long-Term Safety and Efficacy Study of Eszopiclone in Elderly With Primary Chronic Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-904
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Insomnia
Keywords: insomnia; chronic; primary
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Bronchiolitis Obliterans Syndrome | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Week -2 to day 0 single blind one tablet placebo in the evening. Double blind period: Day 1 to Week 12 double blind one tablet placebo in the evening. Follow up period: two weeks (Weeks 13-14) single blind one tablet placebo in evening, and two weeks (Weeks 15-16) no drug washout.
  Interventions: Drug: Placebo
- Eszopiclone (Experimental): Week -2 to day 0 single blind one tablet placebo in evening. Double Blind period: Day 1 to Week 12 double blind one tablet 2 mg of eszopiclone in evening. Follow up period consists of two weeks (Weeks 13-14) single blind one tablet placebo in evening, and two weeks (Weeks 15-16) no drug washout.
  Interventions: Drug: Eszopiclone; Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — 2 mg tablet once per day in the evening
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: Placebo — Tablet one per day in the evening.

SUMMARY:
To evaluate the long-term safety and efficacy of eszopiclone administered for 12 weeks in elderly subjects with primary chronic insomnia.Administration of eszopiclone 2 mg daily at bedtime for 12 weeks in elderly subjects with a diagnosis of primary chronic insomnia will be safe and well tolerated, improve subjective sleep measures, improve measures of Quality of Life and next day insomnia symptoms, and have no significant withdrawal central nervous system adverse events or rebound insomnia.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo controlled, parallel group study of eszopiclone in elderly subjects with primary chronic insomnia. The study will involve up to 9 visits and subject participation will be approximately 18 weeks. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with primary chronic insomnia. Subject is otherwise in good general health, based on screening physical examination and medical history.

Exclusion Criteria:

* Subject has recent history of known clinically significant abnormal laboratory findings.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 388 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, CNS, Study Chair — Sumitomo Pharma America, Inc.
Locations (73):
- United States (73):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Irvine, California
  - La Mesa, California
  - Los Angeles, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Atlanta, Florida
  - Clearwater, Florida
  - Coral Springs, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Gables, Florida
  - Jupiter, Florida
  - Maitland, Florida
  - Naples, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Stockbridge, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Vernon Hills, Illinois
  - Evansville, Indiana
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Braintree, Massachusetts
  - Newton, Massachusetts
  - Florissant, Missouri
  - Hamilton, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Cary, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Mogadore, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Duncansville, Pennsylvania
  - Scotland, Pennsylvania
  - Warwick, Rhode Island
  - Anderson Pharmaceutical Research, Anderson, South Carolina
  - Anderson, South Carolina
  - Simpsonville, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Fairfax, Virginia
  - Richmond, Virginia
  - Spokane, Washington

REFERENCES:
- [Result] Ancoli-Israel S, Krystal AD, McCall WV, Schaefer K, Wilson A, Claus R, Rubens R, Roth T. A 12-week, randomized, double-blind, placebo-controlled study evaluating the effect of eszopiclone 2 mg on sleep/wake function in older adults with primary and comorbid insomnia. Sleep. 2010 Feb;33(2):225-34. doi: 10.1093/sleep/33.2.225. PMID 20175406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 823 participants were screened. Two participants in each arm completed all assessments for the double blind period but discontinued before starting the follow up period (withdrew consent; did not take any single blind medication in follow up period).
Groups:
- Placebo: Placebo tablets
- Eszopiclone: Eszopiclone 2 mg tablets
Period: Double Blind Period
Arm/Group | Placebo | Eszopiclone
Started | 194 | 194
Completed | 148 | 147
Not Completed | 46 | 47
Not completed — Adverse Event | 9 | 14
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Lack of Efficacy | 20 | 11
Not completed — Didnt Meet Entry/Randomization Criteria | 4 | 5
Not completed — Other | 3 | 3
Period: Follow up:2 Week Placebo, 2 Week no Drug
Arm/Group | Placebo | Eszopiclone
Started | 146 (Two subjects withdrew consent prior to starting the follow up period.) | 145 (Two subjects withdrew consent prior to starting the follow up period.)
Completed | 143 | 144
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Eszopiclone | Total
Number analyzed (Participants) | 194 | 194 | 388
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 194 | 194 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (5.2) | 71.6 (5.0) | 72.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 124 | 243
  Male | 75 | 70 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 8 | 17
  White | 181 | 178 | 359
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 194 | 194 | 388
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms/Meters squared] — Body mass index (BMI) is measure of body fat based on height and weight that applies to both adult men and women
  Kilograms/Meters squared | 27.28 (4.98) | 28.25 (4.90) | 27.76 (4.96)
Height [Mean (Standard Deviation); unit: Centimeters] | 165.90 (9.83) | 164.70 (10.04) | 165.30 (9.94)
Weight [Mean (Standard Deviation); unit: kilograms] — Participant Weight in Kilograms
  kilograms | 75.44 (17.07) | 76.98 (16.72) | 76.21 (16.89)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Subject-Reported Total Sleep Time (TST) Averaged Over the 12 Week Double Blind Study Period.
Description: The difference between the total sleep time at baseline and the average total sleep time over the double blind period(average of post-dose values from weeks 3,6,9,12) reported by the participant. The change is calculated as the average over the double blind period minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose)-12 weeks
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment are included. Last Observation Carried Forward. Change calculated as the post-dose measure minus the baseline measure. Number of participants in each arm 194, 194.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 191 | 191
minutes | 33.18 (50.02) | 63.24 (52.76)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

2. Secondary Outcome: Mean Change From Baseline in Subject-reported Total Sleep Time at Various Study Time Points.
Description: The difference between the total sleep time at baseline and at different time points in the double-blind period (weeks 3,6,9,12), the single-blind follow-up (week 14) and the non-drug treatment follow-up (week 16). The change is calculated as the time point value minus the baseline value.
Time Frame: Weeks 0, 3, 6, 9, 12, 14, 16
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment are included. Last Observation Carried Forward. Change calculated as the post-dose measure minus the baseline measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 3 (n=191,190) | 20.65 (42.34) [13.68 to 25.72] | 51.02 (46.43) [44.88 to 56.99]
  Week 6 (n=191,191) | 32.47 (53.31) [25.29 to 39.67] | 61.91 (54.15) [56.18 to 70.63]
  Week 9 (n=191,191) | 38.73 (57.73) [30.99 to 46.75] | 69.00 (61.58) [63.00 to 78.83]
  Week 12 (n=191,191) | 40.86 (60.74) [33.16 to 49.63] | 70.97 (62.18) [64.95 to 81.50]
  Week 14 (n=191,191) | 42.78 (66.52) [35.54 to 53.54] | 50.12 (68.25) [44.83 to 62.92]
  Week 16 (n=191,191) | 37.43 (67.68) [31.36 to 49.07] | 47.17 (63.68) [42.89 to 60.69]

3. Secondary Outcome: Mean Subject-reported Total Sleep Time in Minutes at Various Study Time Points.
Description: The mean total minutes asleep each night at different time points: baseline(week 0), double-blind phase(weeks 3,6,9,12), the single-blind follow-up(week 14),the non-drug treatment follow-up(week 16), and the double-blind average(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0, 3, 6, 9, 12, 14, 16
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment are included. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 0 (n=192,191) | 294.03 (63.30) | 297.86 (56.14)
  Week 3 (n=192,192) | 314.53 (63.52) | 347.37 (57.17)
  Week 6 (n=192,193) | 326.25 (65.41) | 358.72 (61.47)
  Week 9 (n=192,193) | 332.47 (65.25) | 365.80 (64.97)
  Week 12 (n=192,193) | 334.69 (69.91) | 367.75 (66.08)
  Weeks 3,6,9,12 (double blind average)(n=192,193) | 326.98 (62.88) | 360.08 (59.40)
  Week 14 (n=192,193) | 336.55 (71.13) | 347.12 (72.97)
  Week 16 (n=192,193) | 331.29 (72.53) | 344.20 (74.91)

4. Secondary Outcome: Mean Change From Baseline in Subject-reported Sleep Latency (SL) Averaged Over the 12 Week Double Blind Period.
Description: Sleep latency answers how long it takes to fall asleep. The difference between the sleep latency at baseline and the average sleep latency over the double blind period(average of post-dose values from weeks 3,6,9,12) reported by the participant. The change is calculated as the average over the double blind period minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - Week12
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment are included. Last Observation Carried Forward. Number of participants in each arm 194, 194.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 191 | 191
minutes | -19.92 (46.99) | -24.62 (46.32)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0014, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

5. Secondary Outcome: Mean Change From Baseline in Subject-reported Sleep Latency at Various Study Time Points
Description: Sleep latency answers the question: How long did it take you to fall asleep last night? The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 3 (n=191,190) | -13.34 (41.97) [0.78 to 0.90] | -21.89 (44.38) [0.64 to 0.74]
  Week 6 (n=191,191) | -19.69 (52.08) [0.70 to 0.83] | -24.13 (49.20) [0.59 to 0.70]
  Week 9 (n=191,191) | -23.02 (50.75) [0.66 to 0.79] | -24.21 (52.62) [0.57 to 0.68]
  Week 12 (n=191,191) | -23.54 (54.14) [0.64 to 0.78] | -28.35 (49.72) [0.53 to 0.64]
  Week 14 (n=191,191) | -25.08 (58.99) [0.61 to 0.75] | -17.00 (55.55) [0.62 to 0.77]
  Week 16 (n=191,191) | -24.61 (55.22) [0.62 to 0.76] | -18.73 (51.67) [0.60 to 0.74]

6. Secondary Outcome: Mean Subject-reported Sleep Latency Reported at Various Study Time Points.
Description: Sleep latency answers the question: How long did it take you to fall asleep last night? Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the entire double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 0 (n=192,191) | 82.17 (74.08) | 75.68 (56.63)
  Week 3 (n=192,192) | 68.80 (64.51) | 54.69 (46.16)
  Week 6 (n=192,193) | 62.57 (60.06) | 52.11 (48.66)
  Week 9 (n=192,193) | 59.23 (52.05) | 51.75 (51.79)
  Week 12 (n=192,193) | 58.69 (51.84) | 47.66 (39.70)
  Weeks 3,6,9,12 (double blind average)(n=192,193) | 62.32 (54.82) | 51.51 (43.87)
  Week 14 (n=192,193) | 57.23 (49.94) | 58.89 (45.89)
  Week 16 (n=192,193) | 57.62 (51.99) | 57.17 (45.40)

7. Secondary Outcome: Mean Change From Baseline in Subject-reported Wake Time After Sleep Onset (WASO) Averaged Over the 12 Week Double-blind Study Period.
Description: Wake time after sleep onset (WASO) is the time spent awake from sleep onset to final awakening. The difference between WASO at baseline and the average WASO over the double blind period(average of post-dose values from weeks 3,6,9,12). The change is calculated as the average over the double blind period minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) -week 12
Population: Intent to treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment are included. Last observation carried forward (LOCF). Number of participants in each arm 194, 194.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 191
minutes | -14.75 (38.45) | -36.40 (41.29)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

8. Secondary Outcome: Mean Change From Baseline in Subject-reported Wake Time After Sleep Onset (WASO) at Various Study Time Points.
Description: Wake time after sleep onset is the time spent awake from sleep onset to final awakening. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 3 (n=188,190) | -8.55 (35.80) [0.73 to 0.93] | -29.26 (37.68) [0.48 to 0.61]
  Week 6 (n=189,191) | -13.46 (39.01) [0.65 to 0.86] | -36.57 (43.11) [0.39 to 0.51]
  Week 9 (n=189,191) | -17.67 (44.13) [0.57 to 0.77] | -40.32 (45.12) [0.36 to 0.49]
  Week 12 (n=189,191) | -19.13 (43.39) [0.54 to 0.74] | -39.61 (46.48) [0.35 to 0.48]
  Week 14 (n=189,191) | -22.72 (45.00) [0.46 to 0.64] | -32.27 (47.55) [0.39 to 0.55]
  Week 16 (n=189,191) | -20.18 (48.06) [0.45 to 0.64] | -31.13 (51.35) [0.38 to 0.54]

9. Secondary Outcome: Mean Subject-reported Wake Time After Sleep Onset (WASO) at Various Study Time Points
Description: Wake time after sleep onset is the time spent awake from sleep onset to final awakening. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the entire double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 0 (n=190,191) | 90.86 (51.77) | 92.66 (58.11)
  Week 3 (n=190,192) | 83.17 (49.63) | 64.33 (45.97)
  Week 6 (n=192,193) | 77.86 (48.82) | 56.49 (44.25)
  Week 9 (n=192,193) | 73.33 (49.71) | 52.75 (42.51)
  Week 12 (n=192,193) | 72.02 (50.44) | 53.45 (44.23)
  Weeks 3,6,9,12 (double blind average)(n=192,193) | 76.59 (47.52) | 56.68 (42.40)
  Week 14 (n=192,193) | 68.39 (51.87) | 60.71 (47.07)
  Week 16 (n=192,193) | 71.27 (54.61) | 61.84 (48.93)

10. Secondary Outcome: Mean Change From Baseline in Subject-reported Number of Awakenings Averaged Over the 12 Week Double Blind Study Period.
Description: The number of awakenings is the number of times a subject wakes up between the initial onset of sleep and the final awakening. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - Week12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 191
number of awakenings | -0.27 (0.72) | -0.56 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0005, ANCOVA — Multiple comparisons not applied due to only two treatments in study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

11. Secondary Outcome: Mean Change From Baseline in the Number of Subject-reported Awakenings at Various Study Time Points.
Description: The number of awakenings refers to the number of times a subject wakes up between the initial onset of sleep and the final awakening. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
number of awakenings
  Week 3 (n=188,190) | -0.16 (.63) [-0.27 to -0.10] | -0.46 (0.70) [-0.51 to -0.34]
  Week 6 (n=189,191) | -0.24 (0.77) [-0.38 to -0.17] | -0.56 (0.83) [-0.64 to -0.44]
  Week 9 (n=189,191) | -0.33 (0.81) [-0.47 to -0.26] | -0.57 (0.88) [-0.66 to -0.45]
  Week 12 (n=189,191) | -0.35 (0.83) [-0.50 to -0.28] | -0.65 (0.90) [-0.75 to -0.52]
  Week 14 (n=189,191) | -0.38 (0.85) [-0.54 to -0.30] | -0.46 (0.96) [-0.57 to -0.33]
  Week 16 (n=189,191) | -0.35 (0.87) [-0.53 to -0.29] | -0.44 (0.97) [-0.57 to -0.33]

12. Secondary Outcome: Mean Number of Awakenings (Subject-reported) at Various Study Time Points
Description: Number of awakenings is number of times a subject wakes up between initial onset of sleep and final awakening. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
number of awakenings
  Week 0 (n=190,191) | 1.95 (1.00) | 2.10 (1.10)
  Week 3 (n=190,192) | 1.78 (0.91) | 1.66 (0.96)
  Week 6 (n=192,193) | 1.72 (0.93) | 1.55 (1.00)
  Week 9 (n=192,193) | 1.62 (0.94) | 1.54 (1.01)
  Week 12 (n=192,193) | 1.61 (0.94) | 1.46 (1.03)
  Weeks 3,6,9,12 (double blind average)(n=192,193) | 1.68 (0.90) | 1.55 (0.97)
  Week 14 (n=192,193) | 1.58 (0.99) | 1.65 (1.15)
  Week 16 (n=192,193) | 1.61 (0.97) | 1.66 (1.11)

13. Secondary Outcome: Mean Change From Baseline in Subject-reported Quality of Sleep Averaged Over the 12 Week Double Blind Study Period
Description: Quality of sleep was rated by participants on a scale of 0-10, with higher scores representing better quality sleep. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - Week12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 191
units on a scale | 0.68 (1.35) | 1.39 (1.43)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

14. Secondary Outcome: Mean Change From Baseline in Subject-reported Quality of Sleep at Various Study Time Points.
Description: Sleep quality was rated by subjects on a scale from 0-10, with higher scores representing better quality sleep. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=188,190) | 0.37 (0.98) [0.24 to 0.52] | 1.12 (1.18) [0.94 to 1.22]
  Week 6 (n=189,191) | 0.62 (1.31) [0.49 to 0.83] | 1.35 (1.43) [1.16 to 1.50]
  Week 9 (n=189,191) | 0.81 (1.58) [0.68 to 1.06] | 1.52 (1.62) [1.31 to 1.69]
  Week 12 (n=189,191) | 0.92 (1.77) [0.78 to 1.19] | 1.57 (1.73) [1.35 to 1.76]
  Week 14 (n=189,191) | 1.02 (1.88) [0.89 to 1.34] | 1.26 (2.07) [1.03 to 1.48]
  Week 16 (n=189, 191) | 0.88 (1.96) [0.78 to 1.23] | 1.22 (2.06) [1.03 to 1.48]

15. Secondary Outcome: Mean Ratings of Subject-reported Quality of Sleep at Various Study Time Points
Description: Quality of sleep was rated by participants on a scale of 0-10, with higher scores representing better quality sleep. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=190,191) | 4.84 (1.83) | 4.68 (1.94)
  Week 3 (n=190,190) | 5.22 (1.62) | 5.77 (1.82)
  Week 6 (n=192,193) | 5.48 (1.56) | 6.01 (1.77)
  Week 9 (n=192,193) | 5.67 (1.57) | 6.17 (1.71)
  Week 12 (n=192,193) | 5.78 (1.58) | 6.22 (1.70)
  Weeks 3,6,9,12 (double blind average)(n=192, 193) | 5.54 (1.50) | 6.04 (1.68)
  Week 14 (n=192,193) | 5.88 (1.60) | 5.91 (1.76)
  Week 16 (n=192,193) | 5.73 (1.65) | 5.88 (1.75)

16. Secondary Outcome: Mean Change From Baseline in Subject-Reported Depth of Sleep for the Average Reported During the Double-blind Period.
Description: Depth of sleep was reported by study participants using a scale from 0-10, with higher scores representing better sleep. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 188 | 190
units on a scale | 0.69 (1.33) | 1.33 (1.43)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

17. Secondary Outcome: Mean Change From Baseline in Subject-reported Depth of Sleep at Various Study Time Points
Description: Depth of sleep was reported by study participants using a scale from 0-10, with higher scores representing better sleep. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=188, 190) | 0.40 (0.97) | 1.07 (1.16)
  Week 6 (n=189, 191) | 0.62 (1.29) | 1.30 (1.44)
  Week 9 (n=189, 191) | 0.82 (1.54) | 1.46 (1.63)
  Week 12 (n=189, 191) | 0.93 (1.74) | 1.49 (1.73)
  Week 14 (n=189,191) | 1.00 (1.88) | 1.23 (2.08)
  Week 16 (n=189,191) | 0.88 (1.96) | 1.15 (2.05)

18. Secondary Outcome: Mean Subject-reported Depth of Sleep at Various Study Time Points
Description: Depth of sleep was reported by study participants using a scale from 0-10, with higher scores representing better sleep. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=190,191) | 4.87 (1.88) | 4.72 (1.90)
  Week 3 (n=190,192) | 5.29 (1.62) | 5.76 (1.78)
  Week 6 (n=192,193) | 5.51 (1.58) | 6.00 (1.75)
  Week 9 (n=192,193) | 5.71 (1.58) | 6.15 (1.73)
  Week 12 (n=192, 193) | 5.82 (1.59) | 6.18 (1.70)
  Weeks 3,6,9,12 (double blind average)(n=192,193) | 5.58 (1.52) | 6.02 (1.68)
  Week 14 (n=192,193) | 5.89 (1.63) | 5.92 (1.78)
  Week 16 (n=192,193) | 5.76 (1.69) | 5.84 (1.76)

19. Secondary Outcome: Mean Change in Subject-reported Daytime Alertness Averaged Over the 12 Week Double Blind Study Period
Description: Daytime alertness was rated by study participants on a scale of 0-10, with higher scores representing better alertness. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 192
units on a scale | 0.61 (1.30) | 1.02 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

20. Secondary Outcome: Mean Change From Baseline in Subject-reported Daytime Alertness at Various Study Time Points
Description: Daytime alertness was rated by study participants on a scale of 0-10, with higher scores representing better alertness. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=189,191) | 0.39 (0.90) | 0.76 (1.03)
  Week 6 (n=189,192) | 0.55 (1.28) | 0.99 (1.29)
  Week 9 (n=189,192) | 0.72 (1.53) | 1.10 (1.54)
  Week 12 (n=189,192) | 0.78 (1.72) | 1.21 (1.64)
  Week 14 (n=189,192) | 0.85 (1.81) | 1.05 (1.92)
  Week 16 (n=189,192) | 0.78 (1.89) | 0.97 (2.00)

21. Secondary Outcome: Mean Subject-reported Daytime Alertness at Various Study Time Points.
Description: Daytime alertness was rated by study participants on a scale of 0-10, with higher scores representing better alertness. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,193) | 5.34 (1.97) | 5.42 (2.11)
  Week 3 (n=190,191) | 5.74 (1.72) | 6.18 (1.78)
  Week 6 (n=190,192) | 5.89 (1.57) | 6.41 (1.68)
  Week 9 (n=190,192) | 6.06 (1.51) | 6.52 (1.59)
  Week 12 (n=190,192) | 6.13 (1.51) | 6.64 (1.58)
  Weeks 3,6,9,12 (double blind average)(n=190,192) | 5.95 (1.50) | 6.44 (1.59)
  Week 14 (n=190,192) | 6.19 (1.52) | 6.47 (1.63)
  Week 16 (n=190,192) | 6.13 (1.59) | 6.39 (1.60)

22. Secondary Outcome: Mean Change From Baseline in Subject-Reported Ability to Function Averaged Over the 12 Week Double Blind Period
Description: Ability to function was rated by study participants on a scale of 0-10, with higher scores representing better ability to function. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 192
units on a scale | 0.53 (1.29) | 0.91 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

23. Secondary Outcome: Mean Change From Baseline in Subject-reported Ability to Function at Various Study Time Points
Description: Ability to function was rated by study participants on a scale of 0-10, with higher scores representing better ability to function. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=189,191) | 0.36 (0.88) | 0.69 (0.98)
  Week 6 (n=189,192) | 0.46 (1.25) | 0.87 (1.27)
  Week 9 (n=189,192) | 0.62 (1.54) | 0.98 (1.50)
  Week 12 (n=189,192) | 0.69 (1.68) | 1.08 (1.60)
  Week 14 (n=189,192) | 0.75 (1.81) | 0.96 (1.87)
  Week 16 (n=189,192) | 0.69 (1.87) | 0.87 (1.96)

24. Secondary Outcome: Mean Subject-reported Ability to Function at Various Study Time Points
Description: Ability to function was rated by study participants on a scale of 0-10, with higher scores representing better ability to function. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16) & average for double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,193) | 5.62 (2.07) | 5.69 (2.14)
  Week 3 (n=190,191) | 5.98 (1.79) | 6.38 (1.79)
  Week 6 (n=190,192) | 6.09 (1.61) | 6.57 (1.68)
  Week 9 (n=190,192) | 6.24 (1.56) | 6.69 (1.57)
  Week 12 (n=190,192) | 6.32 (1.54) | 6.79 (1.55)
  Weeks 3,6,9,12 (double blind average)(n=190,192) | 6.16 (1.55) | 6.61 (1.59)
  Week 14 (n=190,192) | 6.38 (1.54) | 6.66 (1.57)
  Week 16 (n=190,192) | 6.31 (1.62) | 6.57 (1.57)

25. Secondary Outcome: Mean Change From Baseline in Subject-reported Ability to Concentrate Averaged Over the 12 Week Double Blind Study Period.
Description: Ability to concentrate was rated by study participants on a scale of 0-10, with higher scores representing better concentration. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseliine (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 192
units on a scale | 0.50 (1.30) | 0.96 (1.25)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

26. Secondary Outcome: Mean Change From Baseline in Subject-reported Ability to Concentrate at Various Study Time Points.
Description: Ability to concentrate was rated by study participants on a scale of 0-10, with higher scores representing better concentration. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=189,191) | 0.32 (0.89) | 0.73 (0.96)
  Week 6 (n=189,192) | 0.43 (1.29) | 0.93 (1.24)
  Week 9 (n=189,192) | 0.60 (1.53) | 1.03 (1.48)
  Week 12 (n=189,192) | 0.66 (1.71) | 1.14 (1.57)
  Week 14 (n=189,192) | 0.72 (1.81) | 1.00 (1.87)
  Week 16 (n=189,192) | 0.66 (1.89) | 0.93 (1.93)

27. Secondary Outcome: Mean Subject-reported Ability to Concentrate at Various Study Time Points
Description: Ability to concentrate was rated by study participants on a scale of 0-10, with higher scores representing better concentration. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16) & average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,193) | 5.66 (2.08) | 5.63 (2.15)
  Week 3 (n=190,191) | 5.99 (1.78) | 6.37 (1.80)
  Week 6 (n=190,192) | 6.10 (1.62) | 6.57 (1.69)
  Week 9 (n=190,192) | 6.27 (1.54) | 6.67 (1.58)
  Week 12 (n=190,192) | 6.33 (1.52) | 6.77 (1.57)
  Weeks 3,6,9,12 (double blind average)(n=190,192) | 6.17 (1.54) | 6.60 (1.60)
  Week 14 (n=190,192) | 6.39 (1.53) | 6.64 (1.58)
  Week 16 (n=190,192) | 6.33 (1.61) | 6.56 (1.59)

28. Secondary Outcome: Mean Change From Baseline in Subject-reported Physical Well-Being Averaged Over the 12 Week Double Blind Study Period
Description: Physical well-being was rated by study participants on a scale of 0-10, with higher scores representing better well-being. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 189 | 192
units on a scale | 0.52 (1.28) | 0.87 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

29. Secondary Outcome: Mean Change From Baseline in Subject-reported Physical Well-being at Various Study Time Points.
Description: Physical well-being was rated by study participants on a scale of 0-10, with higher scores representing better well-being. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=189,191) | 0.35 (0.88) | 0.68 (0.99)
  Week 6 (n=189,192) | 0.46 (1.26) | 0.84 (1.27)
  Week 9 (n=189,192) | 0.61 (1.52) | 0.93 (1.51)
  Week 12 (n=189,192) | 0.65 (1.71) | 1.02 (1.62)
  Week 14 (n=189,192) | 0.72 (1.82) | 0.89 (1.92)
  Week 16 (n=189,192) | 0.64 (1.90) | 0.80 (1.97)

30. Secondary Outcome: Mean Subject-reported Physical Well-Being at Various Study Time Points
Description: Physical well-being was rated by study participants on a scale of 0-10, with higher scores representing better well-being. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), & average for double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,193) | 5.45 (1.98) | 5.62 (2.14)
  Week 3 (n=190,191) | 5.80 (1.74) | 6.30 (1.77)
  Week 6 (n=190,192) | 5.92 (1.57) | 6.46 (1.65)
  Week 9 (n=190,192) | 6.06 (1.53) | 6.56 (1.56)
  Week 12 (n=190,192) | 6.11 (1.52) | 6.65 (1.53)
  Weeks 3,6,9,12 (double blind average)(n=190,192) | 5.97 (1.51) | 6.49 (1.56)
  Week 14 (n=190,192) | 6.18 (1.53) | 6.51 (1.56)
  Week 16 (n=190,192) | 6.09 (1.61) | 6.43 (1.56)

31. Secondary Outcome: Mean Change From Baseline in Subject-Reported Counts of Number of Naps Per Week Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the number of naps per week for subjects who napped during the baseline period. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose)- week 12
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment and who napped at baseline are included. Last Observation Carried Forward. Number of participants in each arm 194, 194.
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 110 | 93
number of naps | -0.78 (2.30) | -1.23 (2.11)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.1175, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

32. Secondary Outcome: Mean Change From Baseline In Subject-Reported Counts of Number of Naps Per Week at Various Study Time Points
Description: Change from baseline in the number of naps per week for subjects who napped during the baseline period. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: Intention to Treat (ITT) population; Only subjects in the ITT population with at least one post-dose assessment and who napped at baseline are included. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
number of naps
  Week 3 (n=110,92) | -0.39 (2.04) | -1.15 (2.02)
  Week 6 (n=110,93) | -0.80 (2.49) | -1.26 (2.21)
  Week 9 (n=110, 93) | -0.96 (2.67) | -1.33 (2.51)
  Week 12 (n=110, 93) | -0.96 (2.88) | -1.18 (2.58)
  Week 14 (n=110,93) | -0.71 (2.93) | -1.00 (2.31)
  Week 16 (n=110,93) | -0.92 (2.79) | -1.29 (2.49)

33. Secondary Outcome: Mean Subject-Reported Number of Naps Each Week at Various Study Time Points.
Description: The mean number of naps per week for subjects who napped during the baseline period. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
number of naps
  Week 0 (n=111,94) | 4.03 (4.41) | 3.88 (3.55)
  Week 3 (n=110,92) | 3.67 (4.67) | 2.76 (2.96)
  Week 6 (n=110,93) | 3.26 (4.25) | 2.64 (3.00)
  Week 9 (n=110,93) | 3.10 (4.57) | 2.57 (2.63)
  Week 12 (n=110,93) | 3.10 (5.05) | 2.71 (3.06)
  Weeks 3,6,9,12 (double blind average)(n=110,93) | 3.28 (4.51) | 2.66 (2.74)
  Week 14 (n=110,93) | 3.35 (5.32) | 2.90 (3.12)
  Week 16 (n=110,93) | 3.14 (4.63) | 2.61 (3.15)

34. Secondary Outcome: Mean Change in Subject-Reported Total Nap Time Per Week Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the total time (minutes) spent napping per week for subjects who napped during the baseline period. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 110 | 93
minutes | -36.02 (125.59) | -60.06 (156.49)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0717, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

35. Secondary Outcome: Mean Change From Baseline in Subject-Reported Total Nap Time Per Week at Various Study Time Points.
Description: Change from baseline in the total time (minutes) spent napping per week for subjects who napped during the baseline period. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 3 (n=110,92) | -21.66 (116.53) | -59.06 (158.00)
  Week 6 (n=110,93) | -40.02 (140.47) | -65.99 (163.12)
  Week 9 (n=110,93) | -40.25 (146.42) | -56.59 (184.47)
  Week 12 (n=110,93) | -42.15 (136.85) | -58.22 (163.87)
  Week 14 (n=110,93) | -27.28 (142.36) | -44.48 (165.67)
  Week 16 (n=110,93) | -38.14 (137.69) | -49.15 (202.13)

36. Secondary Outcome: Mean Subject-Reported Total Nap Time at Various Study Time Points
Description: The total time (minutes) spent napping per week for subjects who napped during the baseline period. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
minutes
  Week 0 (n=111,94) | 189.31 (262.08) | 171.62 (237.75)
  Week 3 (n=110,92) | 169.24 (253.66) | 114.43 (151.26)
  Week 6 (n=110,93) | 150.88 (226.90) | 106.99 (133.85)
  Week 9 (n=110,93) | 150.65 (234.11) | 116.39 (156.42)
  Week 12 (n=110,93) | 148.75 (256.87) | 114.76 (149.73)
  Weeks 3,6,9,12 (double blind average)(n=110,93) | 154.88 (237.82) | 112.92 (135.34)
  Week 14 (n=110,93) | 163.61 (274.13) | 128.50 (173.51)
  Week 16 (n=110,93) | 152.76 (246.50) | 123.83 (173.58)

37. Secondary Outcome: Mean Change From Baseline in Subject-Reported Total Nap Time Per Week as a Percent of Total Asleep Time Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the total time spent napping per week stated as a percentage of the total time asleep for subjects who napped during the baseline period. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 110 | 93
percentage of total asleep time | -2.44 (8.29) | -2.98 (5.53)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.1182, ANCOVA — Multiple comparisons not applied due to only two treatments in the study

38. Secondary Outcome: Mean Change From Baseline in Subject-Reported Total Nap Time Stated as a Percentage of the Total Asleep Time at Various Study Time Points
Description: Change from baseline in the total time spent napping per week stated as a percentage of the total time asleep for subjects who napped during the baseline period. The change is calculated as value during double-blind phase(weeks 3,6,9,12), or the single-blind follow-up(week 14), or the non-drug treatment follow-up(week 16) minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
percentage of total asleep time
  Week 3 (n=110,92) | -1.78 (7.00) | -2.77 (5.57)
  Week 6 (n=110,93) | -2.52 (9.09) | -3.16 (5.80)
  Week 9 (n=110,93) | -2.72 (9.26) | -2.94 (6.24)
  Week 12 (n=110,93) | -2.76 (8.98) | -3.04 (5.82)
  Week 14 (n=110,93) | -2.31 (9.22) | -2.14 (5.82)
  Week 16 (n=110,93) | -2.55 (8.62) | -2.38 (6.72)

39. Secondary Outcome: Mean Subject-Reported Total Nap Time Per Week Stated as a Percentage of the Total Asleep Time at Various Study Time Points
Description: Total time spent napping per week stated as a percentage of total time asleep for subjects who napped during baseline period. Mean values reported: baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week14), non-drug treatment follow-up(week 16), & average for double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 32
Measure: Median (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
percentage of total asleep time
  Week 0 (n=111,94) | 9.05 (13.89) | 7.02 (8.34)
  Week 3 (n=110,92) | 7.35 (11.94) | 4.33 (5.53)
  Week 6 (n=110,93) | 6.61 (11.73) | 3.91 (4.83)
  Week 9 (n=110,93) | 6.41 (11.04) | 4.13 (5.15)
  Week 12 (n=110,93) | 6.37 (11.77) | 4.04 (5.00)
  Weeks 3,6,9,12 (double blind average)(n=110,93) | 6.68 (11.37) | 4.09 (4.75)
  Week 14 (n=110,93) | 6.82 (11.17) | 4.93 (6.19)
  Week 16 (n=110,93) | 6.57 (11.00) | 4.69 (6.27)

40. Secondary Outcome: Mean Change From Baseline in Total Sleep Time Measured by Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Participants who wore an actigraph wrist monitor, which monitors rest and activity cycles are included; the resultant data had total sleep time calculated by a Central Reader. The change is calculated as the average over the double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: The subset population wore an actigraph wrist monitor device every day between Weeks -1 and 16. A total of 17 weeks of actigraphy data was collected but only 7 weeks (Weeks 0,1,4,7,12,13,15) of actigraphy data was overread by a Central Reader and had sleep parameters calculated. Last Observation Carried Forward.Actigraphy population N=72,69.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 62 | 61
minutes | 14.40 (38.14) | 17.96 (34.71)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.3010, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

41. Secondary Outcome: Mean Change From Baseline in Total Sleep Time Measured by Actigraphy at Various Study Time Points
Description: Change from baseline in total sleep time for the subset population who wore an actigraph wrist monitor. The actigraph monitors rest and activity cycles; the resultant data had sleep parameters calculated by a Central Reader. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: The subset population wore an actigraph wrist monitor device every day between Weeks -1 and 16. A total of 17 weeks of actigraphy data was collected but only 7 weeks (Weeks 0,1,4,7,12,13,15) of actigraphy data was overread by a Central Reader and had sleep parameters calculated. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 1 (n=60,58) | 3.72 (54.09) | 14.97 (36.91)
  Week 4 (n=61,61) | 17.21 (39.97) | 16.89 (41.00)
  Week 7 (n=62,61) | 15.72 (57.85) | 22.12 (41.02)
  Week 12 (n=62,61) | 18.93 (44.73) | 18.08 (52.57)
  Week 13 (n=62,61) | 15.36 (51.72) | -0.60 (56.17)
  Week 15 (n=62,61) | 13.82 (43.48) | 4.06 (47.60)

42. Secondary Outcome: Mean Total Sleep Time Measured by Actigraphy at Various Study Time Points
Description: Total sleep time for subset who wore actigraph wrist monitor which monitors rest and activity cycles, sleep parameters calculated by Central Reader. Mean values reported:baseline(week0), double-blind(weeks1,4,7,12), single-blind follow-up(week13), non-drug follow-up(week15) & average for double-blind(average of weeks1,4,7,12 values).
Time Frame: Weeks 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 0 (n=64,61) | 351.06 (86.05) | 367.95 (60.86)
  Week 1 (n=64,64) | 354.11 (94.76) | 381.52 (73.83)
  Week 4 (n=67,67) | 366.69 (78.34) | 382.39 (69.41)
  Week 7 (n=68,67) | 368.58 (86.48) | 386.96 (63.89)
  Week 12 (n=68,67) | 368.70 (83.39) | 382.04 (69.98)
  Weeks 1,4,7,12 (double blind average)(n=68,67) | 365.13 (79.31) | 383.30 (63.78)
  Week 13 (n=68,67) | 366.47 (81.33) | 364.87 (74.16)
  Week 15 (n=68,67) | 365.73 (74.47) | 369.23 (64.82)

43. Secondary Outcome: Mean Change From Baseline in Sleep Latency Measured Using Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Sleep latency is the time it takes to fall asleep. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as the average over the double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 62 | 61
minutes | 0.00 (40.75) | 1.47 (26.76)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.7800, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

44. Secondary Outcome: Mean Change From Baseline in Sleep Latency Measured Using Actigraphy at Various Study Time Points
Description: Sleep latency is a measurement of the time it takes to fall asleep. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 1 (n=60,58) | 9.06 (74.76) | -0.25 (18.92)
  Week 4 (n=61,61) | -2.16 (44.61) | -1.48 (27.74)
  Week 7 (n=62,61) | 0.12 (52.95) | -1.62 (26.28)
  Week 12 (n=62,61) | -3.92 (36.22) | 9.34 (57.32)
  Week 13 (n=62,61) | -0.69 (59.32) | 16.13 (66.04)
  Week 15 (n=62,61) | -3.66 (39.21) | 6.44 (36.59)

45. Secondary Outcome: Mean Sleep Latency Values Measured Using Actigraphy at Various Study Time Points.
Description: Sleep latency:measurement of time to fall asleep. Values are for subset who wore an actigraph wrist monitor which monitors rest and activity cycles; sleep parameters calculated by Central Reader.
Time Frame: Weeks 0,1,4,7,12,13,15
Population: The subset population wore an actigraph wrist monitor device every day between Weeks -1 and 16. Mean values reported:baseline(week0), double-blind (weeks 1,4,7,12), single-blind follow-up(week13), non-drug treatment follow-up(week15) & average for double-blind (average of weeks 1,4,7,12 values). Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 0 (n=64,61) | 31.34 (65.06) | 23.89 (24.50)
  Week 1 (n=64,64) | 37.74 (78.14) | 26.72 (36.56)
  Week 4 (n=67,67) | 28.55 (35.46) | 26.62 (43.36)
  Week 7 (n=68,67) | 31.06 (42.82) | 26.89 (33.34)
  Week 12 (n=68,67) | 27.89 (38.78) | 36.93 (57.69)
  Weeks 1,4,7,12 (double blind average)(n=68,67) | 31.20 (36.89) | 29.22 (35.92)
  Week 13 (n=68,67) | 30.40 (41.05) | 43.06 (64.37)
  Week 15 (n=68,67) | 28.80 (37.75) | 34.35 (40.34)

46. Secondary Outcome: Mean Change From Baseline in Wake Time After Sleep Onset (WASO) Measured by Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Wake time after sleep onset is the time spent awake from sleep onset to final awakening. Change is calculated as average over double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 62 | 61
minutes | 4.50 (19.54) | -4.24 (22.91)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0803, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

47. Secondary Outcome: Mean Change From Baseline in Wake Time After Sleep Onset Measured Using Actigraphy at Various Study Time Points
Description: Wake time after sleep onset is the time spent awake from sleep onset to final awakening. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 1 (n=59,58) | 3.17 (16.23) | -6.59 (23.78)
  Week 4 (n=61,61) | 4.67 (23.36) | -3.88 (26.95)
  Week 7 (n=62,61) | 6.57 (30.27) | -4.19 (25.25)
  Week 12 (n=62,61) | 3.24 (17.90) | -2.54 (24.42)
  Week 13 (n=62,61) | 4.98 (22.35) | 0.68 (23.79)
  Week 15 (n=62,61) | 7.74 (25.70) | -0.27 (24.10)

48. Secondary Outcome: Mean Values for Wake Time After Sleep Onset Measured Using Actigraphy at Various Study Time Points
Description: Wake time after sleep onset is time spent awake from sleep onset to final awakening. Mean values reported: baseline(week 0), double-blind phase(weeks 1,4,7,12), single-blind follow-up(week 13), non-drug treatment follow-up(week 15) & average for double-blind phase(average of weeks 1,4,7,12 values).
Time Frame: weeks 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 0 (n=64,61) | 60.27 (29.51) | 63.75 (29.11)
  Week 1 (n=63,64) | 63.53 (31.09) | 55.39 (22.11)
  Week 4 (n=67,67) | 64.16 (32.11) | 58.86 (24.51)
  Week 7 (n=68,67) | 65.81 (35.11) | 58.09 (22.41)
  Week 12 (n=68,67) | 62.41 (30.09) | 60.22 (23.10)
  Weeks 1,4,7,12 (double blind average)(n=68,67) | 63.69 (29.90) | 58.21 (20.76)
  Week 13 (n=68,67) | 64.09 (31.39) | 63.01 (27.84)
  Week 15 (n=68,67) | 67.07 (37.40) | 62.27 (25.77)

49. Secondary Outcome: Mean Change From Baseline in Number of Awakenings Using Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Number of awakenings refers to the number of times a subject awakens between first sleep onset to final awakening. Change is calculated as average over double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 62 | 61
number of awakenings | 0.87 (3.65) | -0.18 (4.28)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.2643, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

50. Secondary Outcome: Mean Change From Baseline in the Number of Awakenings Measured Using Actigraphy at Various Study Time Points.
Description: Number of awakenings refers to the number of times a subject awakens between first sleep onset to final awakening. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
number of awakenings
  Week 1 (n=59,58) | 0.76 (3.09) | -0.54 (4.19)
  Week 4 (n=61,61) | 0.79 (4.62) | 0.04 (5.22)
  Week 7 (n=62,61) | 0.88 (4.73) | -0.21 (5.05)
  Week 12 (n=62,61) | 0.95 (4.60) | -0.10 (4.93)
  Week 13 (n=62,61) | 1.10 (4.69) | 0.01 (4.93)
  Week 15 (n=62,61) | 1.36 (4.35) | -0.13 (5.02)

51. Secondary Outcome: Mean Number of Awakenings Measured Using Actigraphy at Various Study Time Points
Description: Number of awakenings refers to the number of times a subject awakens between first sleep onset to final awakening. Mean values are reported at baseline(week 0), double-blind phase(weeks 1,4,7,12), single-blind follow-up(week 13), non-drug treatment follow-up(week 15), and the average for the double-blind phase(average of weeks 1,4,7,12 values).
Time Frame: Weeks 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
number of awakenings
  Week 0 (n=64,61) | 21.49 (7.53) | 22.84 (6.94)
  Week 1 (n=63,64) | 22.42 (7.17) | 21.86 (5.96)
  Week 4 (n=67,67) | 22.28 (7.30) | 22.51 (6.16)
  Week 7 (n=68,67) | 22.52 (7.93) | 22.19 (6.08)
  Week 12 (n=68,67) | 22.36 (7.76) | 22.37 (6.25)
  Weeks 1,4,7,12 (double blind average)(n=68,67) | 22.40 (7.15) | 22.27 (5.66)
  Week 13 (n=68,67) | 22.55 (7.57) | 22.48 (7.30)
  Week 15 (n=68,67) | 22.87 (7.71) | 22.38 (5.99)

52. Secondary Outcome: Mean Change From Baseline in Number of Naps Per Week Measured Using Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the number of naps per week for subjects who napped during the baseline period. Change is calculated as the average over the double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 58 | 58
number of naps | 1.61 (9.06) | -2.67 (12.61)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0765, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

53. Secondary Outcome: Mean Change From Baseline in the Number of Naps Per Week Measured Using Actigraphy at Various Study Time Points
Description: Change from baseline in the number of naps per week for subjects who napped during the baseline period. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
number of naps
  Week 1 (n=57,55) | 1.33 (9.15) | -0.62 (12.92)
  Week 4 (n=57,58) | 1.02 (11.73) | -3.43 (13.36)
  Week 7 (n=58,58) | 1.68 (10.63) | -2.83 (16.76)
  Week 12 (n=58,58) | 1.86 (9.83) | -3.47 (15.15)
  Week 13 (n=58,58) | 2.73 (10.54) | -4.58 (13.69)
  Week 15 (n=58,58) | 3.41 (11.22) | -0.64 (12.16)

54. Secondary Outcome: Mean Number of Naps Per Week Measured Using Actigraphy at Various Study Time Points
Description: The number of naps per week for subjects who napped during the baseline period. Mean values are reported at baseline(week 0), double-blind phase(weeks 1,4,7,12), single-blind follow-up(week 13), non-drug treatment follow-up(week 15), and the average for the double-blind phase(average of weeks 1,4,7,12 values).
Time Frame: Week 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
number of naps
  Week 0 (n=62,58) | 20.52 (15.63) | 22.33 (15.42)
  Week 1 (n=57,55) | 20.94 (14.99) | 21.69 (15.38)
  Week 4 (n=57,58) | 20.63 (15.38) | 18.90 (13.85)
  Week 7 (n=58,58) | 21.07 (14.93) | 19.50 (15.18)
  Week 12 (n=58,58) | 21.25 (14.29) | 18.86 (15.18)
  Weeks 1,4,7,12 (double blind average)(n=58,58) | 21.01 (13.90) | 19.66 (12.91)
  Week 13 (n=58,58) | 22.12 (15.97) | 17.75 (12.66)
  Week 15 (n=58,58) | 22.80 (15.03) | 21.69 (14.45)

55. Secondary Outcome: Mean Change From Baseline Total Nap Time Per Week Measured by Actigraphy Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the total nap time per week for subjects who napped during the baseline period. Change is calculated as the average over the double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 58 | 58
minutes | 21.26 (196.66) | -40.91 (307.98)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.2967, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

56. Secondary Outcome: Mean Change From Baseline in Total Nap Time Per Week Measured by Actigraphy at Various Study Time Points
Description: Change from baseline in the total nap time per week for subjects who napped during the baseline period. Participants who wore an actigraph wrist monitor to record rest and activity cycles are included; a Central Reader calculated sleep parameters. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 1 (n=57,55) | 2.37 (184.85) | 6.56 (285.45)
  Week 4 (n=57,58) | 6.37 (252.54) | -56.87 (336.01)
  Week 7 (n=58,58) | 23.03 (220.20) | -31.85 (428.85)
  Week 12 (n=58,58) | 38.86 (229.45) | -73.67 (338.69)
  Week 13 (n=58,58) | 64.84 (275.99) | -87.50 (291.01)
  Week 15 (n=58,58) | 61.28 (235.24) | -1.99 (240.85)

57. Secondary Outcome: Mean Total Nap Time Per Week Measured by Actigraphy at Various Study Time Points.
Description: The total nap time per week for subjects who napped during the baseline period. Mean values are reported at baseline(week 0), double-blind phase(weeks 1,4,7,12), single-blind follow-up(week 13), non-drug treatment follow-up(week 15), and the average for the double-blind phase(average of weeks 1,4,7,12 values).
Time Frame: Week 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
minutes
  Week 0 (n=62,58) | 418.49 (368.31) | 438.02 (325.66)
  Week 1 (n=57,55) | 399.19 (298.18) | 445.84 (358.33)
  Week 4 (n=57,58) | 403.18 (328.59) | 381.15 (335.03)
  Week 7 (n=58,58) | 414.68 (315.20) | 406.16 (387.87)
  Week 12 (n=58,58) | 430.50 (313.11) | 364.34 (313.03)
  Weeks 1,4,7,12 (double blind average)(n=58,58) | 412.91 (292.66) | 397.11 (305.65)
  Week 13 (n=58,58) | 456.48 (352.10) | 350.52 (262.61)
  Week 15 (n=58,58) | 452.93 (310.68) | 436.03 (297.32)

58. Secondary Outcome: Mean Change From Baseline in Total Nap Time Per Week as a Percentage of Total Asleep Time Measured by Actigraphy and Averaged Over the 12 Week Double Blind Study Period.
Description: Change from baseline in the total time spent napping per week as a percent of the total time asleep for subjects who napped during the baseline period. Change is calculated as the average over the double blind period (average of post-dose values from weeks 1,4,7,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 58 | 58
percentage of total asleep time | 0.45 (7.84) | -1.75 (8.46)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p = 0.0634, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

59. Secondary Outcome: Mean Change From Baseline in Total Nap Time Per Week as a Percentage of Total Asleep Time as Measured by Actigraphy at Various Study Time Points
Description: Change from baseline in total time spent napping per week as a percent of total time asleep for subjects who napped during the baseline period. Change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 1,4,7,12,13,15
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
percentage of total asleep time
  Week 1 (n=57,55) | 1.38 (13.89) | -0.17 (7.95)
  Week 4 (n=57,58) | -0.56 (8.64) | -2.14 (9.54)
  Week 7 (n=58,58) | 0.18 (9.21) | -1.75 (11.22)
  Week 12 (n=58,58) | 0.46 (7.76) | -2.70 (9.24)
  Week 13 (n=58,58) | 0.94 (7.96) | -2.63 (8.98)
  Week 15 (n=58,58) | 0.95 (8.11) | -0.04 (7.41)

60. Secondary Outcome: Mean Total Nap Time Per Week as a Percentage of Total Asleep Time Measured Using Actigraphy at Various Study Time Points
Description: The total time spent napping per week as a percent of the total time asleep for subjects who napped during the baseline period. Mean values reported: baseline(week 0), double-blind phase(weeks 1,4,7,12), single-blind follow-up(week 13), non-drug treatment follow-up(week 15) & average for double-blind phase(average of weeks 1,4,7,12 values).
Time Frame: Week 0,1,4,7,12,13,15
Population: as for outcome 41
Measure: Median (Standard Deviation); unit: percentage of total asleep time
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 72 | 69
percentage of total asleep time
  Week 0 (n=62,58) | 15.12 (15.32) | 14.05 (9.41)
  Week 1 (n=57,55) | 16.29 (17.55) | 13.89 (10.19)
  Week 4 (n=57,58) | 14.35 (13.63) | 11.92 (9.24)
  Week 7 (n=58,58) | 14.90 (12.97) | 12.30 (10.35)
  Week 12 (n=58,58) | 15.18 (13.23) | 11.36 (9.14)
  Weeks 1,4,7,12 (double blind average)(n=58,58) | 15.16 (12.87) | 12.30 (8.64)
  Week 13 (n=58,58) | 15.66 (13.84) | 11.43 (8.28)
  Week 15 (n=58,58) | 15.66 (12.42) | 14.01 (8.85)

61. Secondary Outcome: Mean Change From Baseline in Insomnia Severity Index Total Score Averaged Over the 12 Week Double Blind Study Period
Description: Change from baseline in the Insomnia Severity Index Total Score which ranges from 0-28. Lower scores represent better sleep. The change is calculated as the average over the double blind period (average of post-dose values from weeks 3,6,9,12) minus the baseline value.
Time Frame: Baseline (week 0), Day 1 (post first dose) - week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 180 | 182
units on a scale | -3.42 (4.38) | -5.67 (5.26)
Statistical Analysis 1: Comparison: Placebo vs Eszopiclone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Multiple comparisons not applied due to only two treatments in the study; ANCOVA with treatment and site type as fixed effects and the baseline as a covariate

62. Secondary Outcome: Mean Change From Baseline in Insomnia Severity Index Total Score at Various Study Time Points
Description: Change from baseline in the Insomnia Severity Index Total Score which ranges from 0-28. Lower scores represent better sleep. The change is calculated as time point value minus the baseline value.
Time Frame: Baseline (week 0), Weeks 3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 3 (n=179,181) | -2.74 (4.51) | -4.94 (5.38)
  Week 6 (n=180,181) | -3.35 (4.89) | -5.67 (5.88)
  Week 9 (n=180,182) | -3.55 (5.10) | -5.89 (5.88)
  Week 12 (n=180,182) | -4.05 (5.15) | -6.18 (5.96)
  Week 14 (n=181,182) | -3.93 (5.25) | -4.06 (5.88)
  Week 16 (n=181,182) | -2.96 (5.16) | -2.96 (5.24)

63. Secondary Outcome: Mean Insomnia Severity Index Total Scores at Various Study Time Points
Description: The Insomnia Severity Index Total Score ranges from 0-28. Lower scores represent better sleep. Mean values are reported at baseline(week 0), double-blind phase(weeks 3,6,9,12), single-blind follow-up(week 14), non-drug treatment follow-up(week 16), and the average for the double-blind phase(average of weeks 3,6,9,12 values).
Time Frame: Weeks 0,3,6,9,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,190) | 16.34 (4.18) | 16.12 (4.81)
  Week 3 (n=180,183) | 13.52 (5.11) | 11.09 (5.48)
  Week 6 (n=181,184) | 12.87 (5.26) | 10.40 (5.87)
  Week 9 (n=181,185) | 12.66 (5.58) | 10.12 (5.77)
  Week 12 (n=181,185) | 12.16 (5.51) | 9.84 (5.63)
  Weeks 3,6,9,12 (double blind average)(n=181,185) | 12.80 (4.87) | 10.36 (5.16)
  Week 14 (n=182,185) | 12.30 (5.68) | 11.94 (5.56)
  Week 16 (n=182,185) | 13.28 (5.39) | 13.05 (5.49)

64. Secondary Outcome: Mean Change From Baseline in Physical Component Summary of the Short Form-36 Scale
Description: Physical component summary of Short Form-36 Scale measures subject's perception of their physical health, where the normal mean for general US population is 50.Scores above/below 50 represent better than/worse than the general US population. Higher scores represent better outcomes. Change is calculated as time point value minus baseline value.
Time Frame: Baseline (week 0), Weeks 6, 12, 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 6 (n=164,165) | 1.01 (7.73) | 1.00 (7.28)
  Week 12 (n=165,166) | 1.38 (7.60) | 1.01 (7.14)
  Week 16 (n=166,166) | 0.69 (7.99) | 0.39 (6.78)

65. Secondary Outcome: Mean Physical Component Summary of the Short Form-36 Scale Scores.
Description: This scale measures subject's perception of their physical health, where the normal mean for general US population is 50.Scores above/below 50 represent better/worse than general US population. Change calculated as time point value minus baseline value: baseline(week0), double-blind (weeks 6,12)and non-drug treatment follow-up(week16).
Time Frame: Weeks 0,6,12,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,190) | 43.99 (10.67) | 45.39 (9.78)
  Week 6 (n=165,168) | 45.06 (10.98) | 46.08 (10.00)
  Week 12 (n=166,169) | 45.38 (10.57) | 46.12 (9.42)
  Week 16 (n=167,169) | 44.70 (10.98) | 45.51 (9.80)

66. Secondary Outcome: Mean Change From Baseline in Mental Component Summary of the Short Form-36 Scale Scores
Description: Mental component summary of Short Form-36 Scale measures subject's perception of their physical health, where the normal mean for general US population is 50. Scores above/below 50 represent better than/worse than the general US population. Higher scores represent better outcomes. Change is calculated as time point value minus baseline value.
Time Frame: Baseline (week 0), Weeks 6,12,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 6 (n=164,165) | -0.44 (7.45) | 0.96 (8.59)
  Week 12 (n=165,166) | -0.94 (8.00) | 0.83 (8.54)
  Week 16 (n=166,166) | -1.22 (8.94) | 0.20 (7.46)

67. Secondary Outcome: Mean Mental Component Summary of the Short Form-36 Scale Scores
Description: This scale measures subject's perception of their physical health, where normal mean for general US population is 50. Scores above/below 50 represent better/worse than general US population. Change calculated: time point value minus baseline value. Mean values: baseline(week0), double-blind phase(weeks 6,12)& non-drug treatment follow-up(week 16).
Time Frame: Weeks 0,6,12,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,190) | 49.69 (9.33) | 49.29 (10.04)
  Week 6 (n=165,168) | 49.49 (10.03) | 49.96 (10.03)
  Week 12 (n=166,169) | 48.98 (10.19) | 49.86 (9.09)
  Week 16 (n=167,169) | 48.68 (10.61) | 49.23 (9.92)

68. Secondary Outcome: Mean Change From Baseline in the Sheehan Disability Scale Total Score.
Description: Sheehan Disability Scale Total Score (range 0-30)measures subject's level of disability & includes: work/school, social life, family life/home responsibilities, days lost &days underproductive; higher scores represent higher degree of disability/impairment. Change is calculated as time point value minus baseline value.
Time Frame: Baseline (week 0), Weeks 6,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 6 (n=164,165) | -2.60 (7.63) | -4.05 (7.42)
  Week 12 (n=165,166) | -3.73 (7.59) | -4.48 (7.72)
  Week 14 (n=166,166) | -3.11 (7.88) | -3.52 (7.15)
  Week 16 (n=166,166) | -3.33 (8.09) | -2.47 (7.14)

69. Secondary Outcome: Mean Sheehan Disability Total Scores
Description: Sheehan Disability Scale Total Score (range 0-30) measures subject's level of disability; includes work/school, social life, family life/home responsibilities, days lost, days underproductive; higher scores represent higher degree of disability/impairment. Mean values reported: baseline, double-blind(weeks 6,12)& follow-up(weeks 14,16).
Time Frame: Weeks 0,6,12,14,16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 194 | 194
units on a scale
  Week 0 (n=192,190) | 11.38 (7.80) | 11.13 (7.63)
  Week 6 (n=165,168) | 8.87 (6.82) | 7.52 (6.81)
  Week 12 (n=166,169) | 7.70 (6.48) | 7.08 (6.85)
  Week 14 (n=166,166) | 8.37 (7.21) | 8.03 (7.10)
  Week 16 (n=167,169) | 8.12 (7.10) | 9.06 (7.71)

ADVERSE EVENTS:
Arm/Group | Placebo | Eszopiclone
Serious Adverse Events (participants affected / at risk) | 2 | 4
Other Adverse Events (participants affected / at risk) | 61 | 86
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Eszopiclone
Appendicitis Perforated (Gastrointestinal disorders) | 1/194 (1) | 0/194 (0)
Cholecystisis (Hepatobiliary disorders) | 0/194 (0) | 1/194 (1)
Pneumonia (Infections and infestations) | 1/194 (1) | 0/194 (0)
Completed Suicide (Psychiatric disorders) | 0/194 (0) | 1/194 (1)
Stress Urinary Incontinence (Renal and urinary disorders) | 0/194 (0) | 1/194 (1)
Rectocele (Reproductive system and breast disorders) | 0/194 (0) | 1/194 (1)
Arteriosclerosis (Vascular disorders) | 0/194 (0) | 1/194 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Eszopiclone
Diarrhoea (Gastrointestinal disorders) | 1/194 (1) | 9/194 (13)
Stomach Discomfort (Gastrointestinal disorders) | 3/194 (7) | 6/194 (7)
Dry Mouth (Gastrointestinal disorders) | 4/194 (4) | 4/194 (5)
Nausea (Gastrointestinal disorders) | 3/194 (6) | 4/194 (4)
Fatigue (General disorders) | 3/194 (3) | 5/194 (5)
Pain (General disorders) | 3/194 (4) | 4/194 (5)
Nasopharyngitis (Infections and infestations) | 12/194 (13) | 11/194 (11)
Influenza (Infections and infestations) | 5/194 (5) | 4/194 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 3/194 (4) | 4/194 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 8/194 (8) | 3/194 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5/194 (6) | 2/194 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/194 (1) | 4/194 (6)
Headache (Nervous system disorders) | 24/194 (45) | 27/194 (51)
Dysgeusia (Nervous system disorders) | 3/194 (4) | 24/194 (35)
Dizziness (Nervous system disorders) | 3/194 (3) | 8/194 (16)
Somnolence (Nervous system disorders) | 4/194 (5) | 5/194 (5)
Anxiety (Psychiatric disorders) | 2/194 (2) | 4/194 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/194 (5) | 5/194 (5)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4/194 (4) | 5/194 (5)
Rash (Skin and subcutaneous tissue disorders) | 4/194 (5) | 2/194 (2)

LIMITATIONS AND CAVEATS:
The data gathered was subjective (except for actigraphy endpoints) and relied either on self reporting or patient assessments derived from standardized questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.